CLINICAL TRIAL: NCT01054157
Title: Expression and Localization of FP Prostaglandin Receptor in Human Ocular Tissues
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: halah el naddaf, meir medical center
Other Study IDs: PROST-1
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Malposition of the Lower Lid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
to approve the expression of PGF2α receptors in hair follicle in ocular skin tissue, explaining the hypertrichotic effect of PG analogues as intraocular pressure lowering treatment.

DETAILED DESCRIPTION:
50 hair follicle dissection - human lower lid skin and lashes will be derived from lateral tarsal strip (LTS) dissected routinely in ectropion repair surgery, the skin strip is dissected routinely in this surgery , without any relation to our study. The study will be planned according to Helsinki declaration for Paraffin embedded LTS tissue sections (4 µ) will be processed and examined in immunohistochemistry lab. FP receptor proteins expression, using subtype-specific polyclonal antibodies, will be detected by the light microscopic level, according to manufacturer instruction.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* malposition of lower eyelid

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: human lower lid skin and lashes will be derived from lateral tarsal strip (LTS) dissected routinely in ectropion repair surgery, the skin strip is dissected routinely in this surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-02

CONTACTS AND LOCATIONS:
Overall Officials: halah el naddaf, doctor, Principal Investigator — Meir Medical Center